CLINICAL TRIAL: NCT06596902
Title: Promoting Physical Activity and Fitness Among Underserved Latino Families Living in U.S.-Mexico Border Regions
Acronym: AFL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Universidad Autonoma de Baja California (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HS-2023-0308; 1R01MD019330-01 (NIH)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Obesity Prevention; Heart Disease
Keywords: Fitness; Healthy Lifestyle; Community Based; Family Program; Latino; U.S.-Mexico Border
MeSH Terms: conditions — Heart Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will test the efficacy and sustainability of an extended, 12-month AFL Program, plus a 12-month active sustainability phase through a two-group parallel arm, cluster randomized controlled trial (RCT) utilizing a Hybrid Type 1 design while also gathering critical information about the implementation process. Participants will be 290 dyads consisting of one parent/caregiver (18 years or older) and one child (6-11 years) from the same household concurrently attending intervention sessions. The child will be the unit of analysis. In each region, 2 of the 4 community centers will be randomized to one of two conditions: 1) a 12-month AFL program or 2) a control group where participants will have access to all recreation center programs available, with exception of the AFL program.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Program (Experimental): The 12-month intervention will progressively increase in intensity & complexity to teach parents/children more complex sports skills & behavioral techniques, & to prepare them to become future team leaders for nutrition education and sports sessions. In addition, the family Olympics events will take place after every 3-month to reinforce progression, social support, & progressive improvements: Phase 1: Beginner (months 0-3) will focus on introductory concepts & basic sports skills & will focus on establishing consistent behavioral patterns & social support. Phase 2: Intermediate (months 4-6) will begin to introduce slightly more complex nutrition & behavioral concepts, increase difficulty of sport skills, & reinforce behavioral patterns from phase 1. Phase 4: Advanced (months 10-12) will teach parents & children advanced sports skills & nutrition knowledge so that they may become team leaders to help implement future activity sessions and nutrition education sessions.
  Interventions: Behavioral: Physical Activity
- Control Group (No Intervention): Centers that are randomly assigned to the control group will continue with regularly schedule programing and activities. Families recruited from control centers will be allowed to take part in all the programs offered at the recreation centers, with exception to the AFL program since it will not be offered at those centers. Control group families will also receive publicly available information regarding the benefits of PA and strategies to become physically active (e.g., CDC PA guidelines websites & handbook). 12-month sustainability phase will involve assessments at the organizational and individual levels. At the organizational level, we will examine the number of AFL sessions held at each recreation center and document the number of phone consultations, length of calls, and barriers addressed. At the individual level, we will examine the number of minutes of adult and child habitual PA.

INTERVENTIONS:
Behavioral: Physical Activity — The 12-month intervention will progressively increase in intensity and complexity to teach parents/children more complex sports skills and behavioral techniques, to prepare them to become future team leaders for nutrition education and sports sessions. In addition, the family Olympics events will take place after every 3-month to reinforce progression, social support; progressive improvements: Phase 1: Beginner (months 0-3) will focus on introductory concepts and basic sports skills and will focus on establishing consistent behavioral patterns and social support. Phase 2: Intermediate (months 4-6) will begin to introduce slightly more complex nutrition behavioral concepts and increase difficulty of sport skills, and reinforce behavioral patterns from phase 1. Phase 4: Advanced (months 10-12) will teach parents and children advanced sports skills ; nutrition knowledge so that they may become team leaders to help implement future activity sessions and nutrition education sessions.
  Arms: Intervention Program

SUMMARY:
This study has the goal to increase physical activity and fitness among Latinos in San Diego, California and Mexicali, Baja California (U.S.-Mexico border) since these cities have similar diseases such as high rates of heart disease and obesity. Therefore there is a need to have physical activity programs for children and their families. We will collaborate with community centers to have this program available.

DETAILED DESCRIPTION:
The U.S. and Mexico share similar population disease patterns such as high rates of chronic diseases (e.g.,heart disease and obesity). Individuals residing in border regions often travel back and forth between the U.S. and Mexico, which exposes them to both different and similar obesogenic, socio-cultural, and physical environments. This frequent transnational interaction has led researchers to classify border cities as one region that should be studied as a whole. As such, it is important to systematically study border populations and develop effective interventions and public policy for this region. This study will test the efficacy and sustainability of a 12-month family-centered behavioral cluster randomized intervention, Athletes for Life (AFL), plus a 1-year active sustainability phase in community recreation centers in San Diego, California (U.S.) and Mexicali, Baja California (Mexico). This study will also assess intervention implementation outcomes, including program acceptability and feasibility by families and community recreation center staff. A total of 8 community recreation centers and 290 parent/child dyads (4 in San Diego and 4 in Mexicali) will be randomized to either a control group consisting of standard recreation center classes (delivered by regular recreation center staff) or an experimental group consisting of the multilevel AFL behavioral intervention (delivered by study staff). This study aims to increase total habitual physical activity (PA) and cardiovascular fitness (CVF) in a U.S.-Mexico transborder population that experiences disproportionately high rates of obesity. We will harness our research team's extensive experience in developing multi-level interventions to promote behavior change among Latinos, and leverage a strong community-academic collaboration that maximizes community impact and sustainability. The long-term goal of this project is to reduce cardiovascular disease and cardiometabolic risk factors among underserved children and their families in the US-Mexico border region. This research will provide novel empirical evidence for the efficacy, scalability, and sustainability of a multilevel fitness- and lifestyle-oriented family approach delivered in collaboration with community centers among underserved Latino families in the U.S.-Mexico border region.

ELIGIBILITY:
Inclusion Criteria:

* parents aged ≥18 years
* children aged 6-11 years
* living in the target community (within 5 miles of one of targeted community centers)

Exclusion Criteria:

* for the parent or child are presence of a medical or physical condition that is contraindicated to participating in sports/exercise (e.g., negative score on the Physical Activity Readiness Questionnaire (PAR-Q)).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Child Physical Activity (PA) | 1 year
  Total PA (mean minutes/day) in children will be measured objectively with a wrist-worn ActiGraph GT9X Link (Pensacola, United States). According to recommended procedures[84], children will be asked to wear the accelerometer continuously on their non-preferred wrist for seven days. Parents will be provided with a sleep diary where they will record their child's wake/sleep times and periods of non-wear. Child and adult CVF performance will be measured via the 1-mile run/walk time in seconds at a local park (usually adjacent to the Community Centers). Study staff will utilize stop watches to collect total mile run time in seconds and record the time in each participant's record log. In addition, a measurement staff will run/walk along with each child participant and provide them with verbal encouragement to put forth their best effort.

SECONDARY OUTCOMES:
Implementation | 1 year
  Will be assessed at multiple levels: participant/families, research team (including Promotores), and Community Center staff. At the participant level, parent-child focus groups will be held and anonymous surveys to assess program satisfaction will be administered. At the staff level; staff and students will be evaluated every 3 months for fidelity by the intervention coordinator through checklists and weekly logs, as well as surveys assessing the feasibility of the program. At the community center level; they will complete brief online surveys involving policy implications, program feasibility, intervention adoption and costs, and reach of recruitment and outreach efforts. Additionally, phone interviews will be held by study personnel to assess appropriateness and sustainability of the AFL intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noe C Crespo, MS, MPH, PhD, Principal Investigator — San Diego State University; Daniela G Gonzalez-Valencia, PhD, Principal Investigator — Universidad Autonoma de Baja California
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be analyzed for the study primary and secondary outcomes. IPD may be shared according to NIH and institutional policies.